CLINICAL TRIAL: NCT04741542
Title: Phase 1, Open-Label, Dose Escalation Study to Assess the Safety of SP-420 in the Treatment of Transfusional Iron Overload
Brief Title: Safety of SP-420 in the Treatment of Transfusional Iron Overload
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is on hold by FDA in the US.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Abfero Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 20-0138; HSC20210039H (Other: UT Health Science Center San Antonio)
Record Dates: First submitted 2021-01-19; First posted 2021-02-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Iron Overload
MeSH Terms: conditions — Iron Overload | interventions — SP-420

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Study subjects will receive a 14mg/kg starting dose of SP-420 three times a week
  Interventions: Drug: SP-420
- Group B (Experimental): Study subjects will receive a 28mg/kg starting dose of SP-420 three times a week
  Interventions: Drug: SP-420
- Group C (Experimental): Study subjects will receive a 42mg/kg starting dose of SP-420 three times a week
  Interventions: Drug: SP-420
- Group D (Experimental): Study subjects will receive a 56mg/kg starting dose of SP-420 three times a week
  Interventions: Drug: SP-420

INTERVENTIONS:
Drug: SP-420 — This study aims to establish the safety of SP-420 administered orally three times per week (TIW).
  Other Names: (4S)-4,5-dihydro-2-[2-hydroxy-4-[2-(2-methoxyethoxy)ethoxy]phenyl]-4-methyl-4-thiazolecarboxylic acid

SUMMARY:
This study enrolls patients with myelodysplastic syndrome (MDS) and myelofibrosis (MFS), with transfusional iron overload and treats them with the investigational iron chelator, SP-420. SP-420 may be better tolerated and safer than commercially available iron chelators. Iron chelation therapy (ICT) has been shown to improve outcomes in iron overload, but adherence is poor due to problems related to ease of administration, tolerability, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Diagnosis of MDS or MF with transfusional iron overload
3. Patients with MDS, will include only those with MDS Revised international prognostic scoring system (IPSS-R) risk group of intermediate, high, or very high.
4. Patients with MF, will include only those with Dynamic International Prognostic Scoring System-Plus (DIPSS=Plus) risk category of intermediate-1, intermediate-2, and high risk.
5. Patients with sickle cell disease and transfusional iron overload
6. Not appropriate for other iron chelation therapy, per physician
7. Received 10 or more units of packed red blood cells in the preceding 24 months and remains red cell transfusion dependent
8. ECOG ≤ 3
9. ALT ≤ 3 times the upper limit of the normal range
10. Estimate glomerular filtration rate calculated using Cockroft Gault of ≥ 60 mL/min/1.73m2
11. Serum ferritin ≥1000 ng/ml
12. Willing to comply with all study procedures and be available for the duration of the study
13. Able to take oral medication and be willing to adhere to study medication for 28 days
14. Female patient must be post-menopausal (no menses for > 12 consecutive months) or surgically sterile (i.e., bilateral oophorectomy, hysterectomy, or tubal sterilization; must agree to completely abstain for heterosexual intercourse; or, if sexually active, must agree to use 1 of the following methods for birth control from the date she signs the consent form until 30 days after final dose of the study drug.

    * Progesterone implant
    * Intrauterine device
    * Combination of 2 highly effective birth control methods (e.g., diaphragm/or cervical cap with spermicide plus a condom, hormonal contraception plus a barrier method, partner with vasectomy conducted >60 days before screening visit plus a hormone or barrier method
15. Male patients must agree to use 1 of the following methods for birth control from the date he signs the consent form until 30 days after final dose of the study drug: be surgically sterile by vasectomy conducted > 60 days before screening visit plus use a barrier method, or, must agree to completely abstain from heterosexual intercourse, or must agree to use a combination of 2 highly effective birth control methods (e.g., diaphragm/or cervical cap with spermicide plus a condom, hormonal contraception plus a barrier method), or have a post-menopausal partner plus barrier method.

Exclusion Criteria:

1. History of kidney disease including the renal Fanconi syndrome
2. Proteinuria on urine dipstick greater than trace positive
3. Pregnant, intending to become pregnant during the study, or breastfeeding
4. Receiving another investigational drug within 30 days or 3 half-lives of the discontinued investigational agent, whichever is greater, of signing consent
5. History of significant hepatic impairment, defined by Child-Pugh class C
6. Active hepatitis B or C disease, evidenced by positive viral PCR
7. Symptomatic heart failure
8. Receiving active cytotoxic chemotherapy or radiation therapy for a second malignancy (hormonal therapy or topical therapy for squamous cell/basal cell cutaneous tumors are allowed). Treatment of the underlying hematologic malignancy with azacytidine, decitabine, venetoclax, lenalidomide, or ruxolitinib is permitted. Treatment with the supportive care agents luspatercept or erythropoietin agonists is permitted.
9. Concurrent treatment with Exjade/Jadenu (deferasirox), Desferal (deferoxamine), or Ferriprox (deferiprone) are not permitted. Patients are allowed to stop these chelators and participate in this trial 14 days after discontinuation of the other chelator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 28 Days
  Count of adverse events induced by SP-420
Completion at original dose | 28 Days
  Number of subjects that completed the study at the original starting dose of that group

CONTACTS AND LOCATIONS:
Overall Officials: Supreet Kaur, MD, Principal Investigator — UT Health San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided